CLINICAL TRIAL: NCT02899494
Title: Effect of the "Adjusted Vocal Expression" Method on the Satisfaction of Parturients About Their Childbirth (NaîtreEnchanté)
Brief Title: Effect of the "Adjusted Vocal Expression" Method on the Satisfaction of Parturients About Their Childbirth
Acronym: NaitreEnchan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2012/10; 2012-A00716-37 (Other: ANSM)
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Pregnancy
MeSH Terms: interventions — Prenatal Education; Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Antenatal classes
  Interventions: Other: Antenatal classes
- Group B (Experimental): Physical and psychic preparation
  Interventions: Other: Physical and psychic preparation

INTERVENTIONS:
Other: Antenatal classes
  Arms: Group A
Other: Physical and psychic preparation
  Arms: Group B

SUMMARY:
To emit voluntarily sounds mastered during the childbirth is a practice found in certain cultures of country of Africa or Muslim or gypsy traditions. Today, because of the medical coverage and because of the childbirth in a hospital environment, this tradition is not anymore transmitted.

The emission of a sound vibration conjugated to a positive intention managed during the childbirth was experimented with around thirty mothers. In the term of this pilot study, most of the women expressed one felt very positive towards the new method, in particular when they compared it with a previous childbirth where this method was not used.

During these childbirths, the midwives also indicated a shortening of the working time.

The present study aim essentially is to confirm the positive effect of the method on the felt of the childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Women of more than 18 years old
* Primipara
* Patients joining the antenatal classes dispensed by the midwives.
* Patients affiliated to a national insurance scheme or benefiting from such a diet
* Patients having given a written consent form

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-11-07 (Actual); Study Completion 2016-11-07 (Actual)

PRIMARY OUTCOMES:
Childbirth Perception Questionnaire (CPQ) score | 5 months
  French adaptation of CPQ score

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc AYOUBI, PhD, Principal Investigator — Hopital Foch
Locations (2):
- France (2):
  - Maternité Catherine BARET de Pertuis, Pertuis
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No